CLINICAL TRIAL: NCT01227187
Title: Safety and Dose Finding Study of Xigris (Drotrecogin Alfa Activated) as an Anti-coagulant in End Stage Renal Disease (ESRD) Patients Treated With Hemodialysis (HD)
Brief Title: Safety and Dose Finding Study of Xigris in Hemodialysis Patients
Acronym: Xigris1003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Mardi Gomberg -Maitland, Professor, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F1K-MC-1003
Record Dates: First submitted 2010-07-14; First posted 2010-10-25 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2020-11

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Anticoagulation; Xigris; PTT
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — drotrecogin alfa activated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xigris (Experimental): Drotrecogin alfa activated (Xigris) used as anticoagulant in patients treated with hemodialysis.
  Interventions: Drug: Drotrecogin alfa activated (Xigris)

INTERVENTIONS:
Drug: Drotrecogin alfa activated (Xigris) — We will test different dose regimens of Drotrecogin alfa activated (Xigris) to determine the optimal dose to achieve PTT between 65 and 100 secs. The initial patients will receive Xigris dosed at an infusion rate of 12 mcg/kg/h via pre-filter arterial drip chamber via a standard IV pump. The PTT will be assessed at baseline,15,30,60,120 and 180 mins. Xigris dose will be adjusted in the following patients if the afferent PTT rises above 100 secs (normal range 25-40 secs) or if PTT remains <65 secs. If PTT remains less than 65 secs, the dose will be increased to the second dose regiment of 18 mcg/kg/hr. The dose escalation will continue in increments of 6 mcg/kg/h to a maximum dose of 36 mcg/kg/h. Each patient will receive Xigris only once.
  Other Names: Drotrecogin alfa (activated)

SUMMARY:
The purpose of the study is to assess the safety of Xigris (Drotrecogin alfa) as an anticoagulant at different dose levels during dialysis treatment in patients with End Stage Renal Disease (ESRD).

DETAILED DESCRIPTION:
In United States, there are over 300,000 patients with ESRD who require hemodialysis. Clinical hemodialysis takes place three times a week and is dependent on adequate anticoagulation throughout the three to four hour procedure. Infection is one of the most common causes of death for patients with ESRD treated with hemodialysis (25%).

Xigris (drotrecogin alfa activated) is a recombinant form of human activated protein C and is successfully used for treatment of adult patients with severe sepsis. In addition to its fibrinolytic properties, drotrecogin alpha has both an anti-inflammatory effect, and an anti-coagulant effect. However, there are few safety and no efficacy data on the effect of Xigris in ESRD patients as an anticoagulant.

ELIGIBILITY:
Inclusion Criteria:

1. >18
2. Usually used heparin with HD

Exclusion Criteria:

1. Plt <100
2. Pregnancy
3. H/o bleeding diathesis
4. H/o CVA
5. Pt on Ticlid/plavix/warfarin
6. SBP >200
7. BASELINE PTT>50
8. INR>1.6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakhmir S Chawla, MD, Principal Investigator — George Washington University
Locations (1):
- The George Washington University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Hakim RM, Held PJ, Stannard DC, Wolfe RA, Port FK, Daugirdas JT, Agodoa L. Effect of the dialysis membrane on mortality of chronic hemodialysis patients. Kidney Int. 1996 Aug;50(2):566-70. doi: 10.1038/ki.1996.350. PMID 8840287
- [Background] Hakim RM, Breyer J, Ismail N, Schulman G. Effects of dose of dialysis on morbidity and mortality. Am J Kidney Dis. 1994 May;23(5):661-9. doi: 10.1016/s0272-6386(12)70276-7. PMID 8172208
- [Background] Held PJ, Port FK, Webb RL, Wolfe RA, Bloembergen WE, Turenne MN, Holzman E, Ojo AO, Young EW, Mauger EA, et al. Excerpts from United States Renal Data System 1995 Annual Data Report. Am J Kidney Dis. 1995 Oct;26(4 Suppl 2):S1-186. No abstract available. PMID 7573030
- [Background] Held PJ, Port FK, Wolfe RA, Stannard DC, Carroll CE, Daugirdas JT, Bloembergen WE, Greer JW, Hakim RM. The dose of hemodialysis and patient mortality. Kidney Int. 1996 Aug;50(2):550-6. doi: 10.1038/ki.1996.348. PMID 8840285
- [Background] Kimmel PL, Peterson RA, Weihs KL, Simmens SJ, Alleyne S, Cruz I, Veis JH. Psychosocial factors, behavioral compliance and survival in urban hemodialysis patients. Kidney Int. 1998 Jul;54(1):245-54. doi: 10.1046/j.1523-1755.1998.00989.x. PMID 9648085
- [Background] Lowrie EG, Laird NM, Parker TF, Sargent JA. Effect of the hemodialysis prescription on patient morbidity: report from the National Cooperative Dialysis Study. N Engl J Med. 1981 Nov 12;305(20):1176-81. doi: 10.1056/NEJM198111123052003. PMID 7027040
- [Background] Lowrie EG, Lew NL. Death risk in hemodialysis patients: the predictive value of commonly measured variables and an evaluation of death rate differences between facilities. Am J Kidney Dis. 1990 May;15(5):458-82. doi: 10.1016/s0272-6386(12)70364-5. PMID 2333868
- [Background] Owen WF Jr, Lew NL, Liu Y, Lowrie EG, Lazarus JM. The urea reduction ratio and serum albumin concentration as predictors of mortality in patients undergoing hemodialysis. N Engl J Med. 1993 Sep 30;329(14):1001-6. doi: 10.1056/NEJM199309303291404. PMID 8366899
- [Background] Causes of death. USRDS. United States Renal Data System. Am J Kidney Dis. 1997 Aug;30(2 Suppl 1):S107-17. No abstract available. PMID 9259696
- [Background] Kimmel PL, Phillips TM, Simmens SJ, Peterson RA, Weihs KL, Alleyne S, Cruz I, Yanovski JA, Veis JH. Immunologic function and survival in hemodialysis patients. Kidney Int. 1998 Jul;54(1):236-44. doi: 10.1046/j.1523-1755.1998.00981.x. PMID 9648084
- [Background] Yeun JY, Levine RA, Mantadilok V, Kaysen GA. C-Reactive protein predicts all-cause and cardiovascular mortality in hemodialysis patients. Am J Kidney Dis. 2000 Mar;35(3):469-76. doi: 10.1016/s0272-6386(00)70200-9. PMID 10692273
- [Background] Kaysen GA. Biological basis of hypoalbuminemia in ESRD. J Am Soc Nephrol. 1998 Dec;9(12):2368-76. doi: 10.1681/ASN.V9122368. PMID 9848794
- [Background] Patient mortality and survival. USRDS. United State Renal Data System. Am J Kidney Dis. 1997 Aug;30(2 Suppl 1):S86-106. No abstract available. PMID 9259695
- [Background] Kaysen GA. Role of inflammation and its treatment in ESRD patients. Blood Purif. 2002;20(1):70-80. doi: 10.1159/000046988. PMID 11803162
- [Background] Bologa RM, Levine DM, Parker TS, Cheigh JS, Serur D, Stenzel KH, Rubin AL. Interleukin-6 predicts hypoalbuminemia, hypocholesterolemia, and mortality in hemodialysis patients. Am J Kidney Dis. 1998 Jul;32(1):107-14. doi: 10.1053/ajkd.1998.v32.pm9669431.
- [Background] Kaysen GA. C-reactive protein: a story half told. Semin Dial. 2000 May-Jun;13(3):143-6. doi: 10.1046/j.1525-139x.2000.00038.x. No abstract available. PMID 10833771
- [Background] Owen WF, Lowrie EG. C-reactive protein as an outcome predictor for maintenance hemodialysis patients. Kidney Int. 1998 Aug;54(2):627-36. doi: 10.1046/j.1523-1755.1998.00032.x. PMID 9690231
- [Background] Bleyer AJ, Russell GB, Satko SG. Sudden and cardiac death rates in hemodialysis patients. Kidney Int. 1999 Apr;55(4):1553-9. doi: 10.1046/j.1523-1755.1999.00391.x. PMID 10201022
- [Background] Bernard GR, Vincent JL, Laterre PF, LaRosa SP, Dhainaut JF, Lopez-Rodriguez A, Steingrub JS, Garber GE, Helterbrand JD, Ely EW, Fisher CJ Jr; Recombinant human protein C Worldwide Evaluation in Severe Sepsis (PROWESS) study group. Efficacy and safety of recombinant human activated protein C for severe sepsis. N Engl J Med. 2001 Mar 8;344(10):699-709. doi: 10.1056/NEJM200103083441001. PMID 11236773
- [Background] Bernard GR, Ely EW, Wright TJ, Fraiz J, Stasek JE Jr, Russell JA, Mayers I, Rosenfeld BA, Morris PE, Yan SB, Helterbrand JD. Safety and dose relationship of recombinant human activated protein C for coagulopathy in severe sepsis. Crit Care Med. 2001 Nov;29(11):2051-9. doi: 10.1097/00003246-200111000-00003. PMID 11700394
- [Background] Bernard GR, Macias WL, Joyce DE, Williams MD, Bailey J, Vincent JL. Safety assessment of drotrecogin alfa (activated) in the treatment of adult patients with severe sepsis. Crit Care. 2003 Apr;7(2):155-63. doi: 10.1186/cc2167. Epub 2003 Feb 28. PMID 12720562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted on stable inpatient HD patients between October 2008 and September 2010. The study design was based on different possible dose levels of APC infusion: 12, 18, 24, 30 μg/kg/h. The initial starting dose of APC for the first patient was 12 μg/kg/h. When a study patient's PTT was <60 s, the starting dose for the next study patient was increased by 6. There were no patient's in the 30 μg/kg/h group with a PTT of <60 s
Pre-assignment Details: Participants were evaluated for inclusion and exclusion criteria and immediately enrolled in the study.
Groups:
- APC Initiation Dose of 12 μg/kg/h: Activated protein C initiation dose of 12 μg/kg/h for the first patient
- APC Initiation Dose of 18 μg/kg/h: Activated protein C initiation dose of 18 μg/kg/h
- APC Initiation Dose of 24 μg/kg/h: Activated protein C initiation dose of 24 μg/kg/h
- APC Initiation Dose of 30 μg/kg/h: Activated protein C initiation dose of 30 μg/kg/h
Period: Overall Study
Arm/Group | APC Initiation Dose of 12 μg/kg/h | APC Initiation Dose of 18 μg/kg/h | APC Initiation Dose of 24 μg/kg/h | APC Initiation Dose of 30 μg/kg/h
Started | 1 | 3 | 3 | 5
Completed | 1 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infusion Rate of 12 mcg/kg/h | Infusion Rate of 18 mcg/kg/h | Infusion Rate of 24 mcg/kg/h | Infusion Rate of 30 mcg/kg/h | Total
Number analyzed (Participants) | 1 | 3 | 3 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (0) | 46 (21.3) | 48.7 (13.1) | 53.2 (7.9) | 49 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 0 | 2 | 2 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 1 | 0 | 1 | 2
  Black | 1 | 2 | 3 | 4 | 10
Height [Mean (Standard Deviation); unit: inches] | 66 (0) | 68.7 (2.9) | 73.3 (5.1) | 68.8 (4.1) | 69.7 (4.2)
Weight [Mean (Standard Deviation); unit: kilograms] | 96 (00) | 69.6 (17.6) | 104.5 (12.6) | 79.4 (29.8) | 84.6 (29.7)
Diabetes [Count of Participants; unit: Participants] | 0 | 0 | 3 | 3 | 6
Congestive heart failure [Count of Participants; unit: Participants] | 0 | 0 | 1 | 2 | 3
WBC [Mean (Standard Deviation); unit: 10^3/µL] | 6.0 (0) | 5.9 (1.8) | 8.1 (0.7) | 6.4 (1.2) | 6.7 (1.4)
Red blood cells [Mean (Standard Deviation); unit: million/mm^3] | 3.6 (0) | 2.7 (0.4) | 3.4 (0.9) | 3.2 (0.5) | 3.1 (0.6)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 9.9 (0) | 7.2 (0.6) | 9.9 (1.4) | 9.0 (1.4) | 9.0 (1.0)
Hematocrit [Mean (Standard Deviation); unit: Percentage of red blood cells in blood] | 31.2 (0) | 23.2 (2.5) | 30.9 (4.0) | 27.9 (3.6) | 27.8 (3.6)
Platelets [Mean (Standard Deviation); unit: 10^9 per liter] | 333 (0) | 196.7 (113.7) | 315 (82.3) | 220.2 (84.5) | 247.4 (95.5)
BUN [Mean (Standard Deviation); unit: mg/dL] | 26 (0) | 36.3 (9.5) | 47 (17.4) | 53.2 (17.1) | 45.2 (17.1)
Creatinine [Mean (Standard Deviation); unit: μmol/L] | 15 (0) | 7.8 (1.1) | 7.8 (0.5) | 9.2 (3.6) | 9.0 (3.0)
Prothrombin time [Mean (Standard Deviation); unit: seconds] | 13.2 (0) | 14.6 (0.2) | 14.2 (1.0) | 13.1 (1.0) | 13.8 (1.0)
Partial thromboplastin time [Mean (Standard Deviation); unit: Seconds] | 38.1 (0) | 37.3 (4.3) | 37.6 (1.3) | 35.5 (6.1) | 36.7 (4.3)
International Normalized Ratio [Mean (Standard Deviation); unit: Ratio] | 1.1 (0) | 1.2 (0.1) | 1.2 (0.2) | 1.0 (0.1) | 1.1 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Partial Thromboplastin Time (PTT) at 15 Minutes
Description: PTT level during a hemodialysis treatment will be used to assess the effectiveness of Xigris as an anticoagulant.
Time Frame: PTT level at 15 minutes after start up of Xigris during the hemodialysis treatment.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- APC Initiation Dose 12 μg/kg/h: APC Initiation dose 12 μg/kg/h
- APC Initiation Dose 18 μg/kg/h: APC Initiation dose 18 μg/kg/h
- APC Initiation Dose 24 μg/kg/h: APC Initiation dose 24 μg/kg/h
- APC Initiation Dose 30 μg/kg/h: APC Initiation dose 30 μg/kg/h
Arm/Group | APC Initiation Dose 12 μg/kg/h | APC Initiation Dose 18 μg/kg/h | APC Initiation Dose 24 μg/kg/h | APC Initiation Dose 30 μg/kg/h
Number analyzed (Participants) | 1 | 3 | 3 | 5
Seconds | 38.4 (NA) — Only 1 subject in arm | 38.4 (4.6) | 45.4 (5.1) | 49.7 (12.0)

2. Primary Outcome: Mean Partial Thromboplastin Time (PTT) at 30 Minutes
Description: PTT level during a hemodialysis treatment will be used to assess the effectiveness of Xigris as an anticoagulant.
Time Frame: PTT level at 30 minutes after start up of Xigris during the hemodialysis treatment.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | APC Initiation Dose 12 μg/kg/h | APC Initiation Dose 18 μg/kg/h | APC Initiation Dose 24 μg/kg/h | APC Initiation Dose 30 μg/kg/h
Number analyzed (Participants) | 1 | 3 | 3 | 5
Seconds | 36.2 (NA) — Only 1 subject in arm | 35.7 (3.4) | 48.2 (8.8) | 51.3 (12.0)

3. Primary Outcome: Mean Partial Thromboplastin Time (PTT) at 60 Minutes
Description: PTT level during a hemodialysis treatment will be used to assess the effectiveness of Xigris as an anticoagulant.
Time Frame: PTT level at 60 minutes after start up of Xigris during the hemodialysis treatment.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | APC Initiation Dose 12 μg/kg/h | APC Initiation Dose 18 μg/kg/h | APC Initiation Dose 24 μg/kg/h | APC Initiation Dose 30 μg/kg/h
Number analyzed (Participants) | 1 | 3 | 3 | 5
Seconds | 39.8 (NA) — Only 1 subject in arm | 36.4 (1.4) | 39.2 (8.0) | 52.6 (16.1)

4. Primary Outcome: Mean Partial Thromboplastin Time (PTT) at 120 Minutes
Description: PTT level during a hemodialysis treatment will be used to assess the effectiveness of Xigris as an anticoagulant.
Time Frame: PTT level at 120 minutes after start up of Xigris during the hemodialysis treatment.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | APC Initiation Dose 12 μg/kg/h | APC Initiation Dose 18 μg/kg/h | APC Initiation Dose 24 μg/kg/h | APC Initiation Dose 30 μg/kg/h
Number analyzed (Participants) | 1 | 3 | 3 | 4
Seconds | 39.4 (NA) — Only one subject in arm. | 42.8 (4.6) | 51.2 (7.8) | 54.1 (14.2)

5. Primary Outcome: Mean Partial Thromboplastin Time (PTT) at 180 Minutes
Description: PTT level during a hemodialysis treatment will be used to assess the effectiveness of Xigris as an anticoagulant.
Time Frame: PTT level at 180 minutes after start up of Xigris during the hemodialysis treatment.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | APC Initiation Dose 12 μg/kg/h | APC Initiation Dose 18 μg/kg/h | APC Initiation Dose 24 μg/kg/h | APC Initiation Dose 30 μg/kg/h
Number analyzed (Participants) | 1 | 3 | 3 | 4
Seconds | 35.6 (NA) — Only 1 subject in arm | 40.9 (1.8) | 44.5 (11.1) | 52.4 (13.3)

ADVERSE EVENTS:
Time Frame: Enrollment until post-treatment day 14
Arm/Group | APC Initiation Dose 12 μg/kg/h | APC Initiation Dose 18 μg/kg/h | APC Initiation Dose 24 μg/kg/h | APC Initiation Dose 30 μg/kg/h
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/3 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APC Initiation Dose 12 μg/kg/h (N=1) | APC Initiation Dose 18 μg/kg/h (N=3) | APC Initiation Dose 24 μg/kg/h (N=3) | APC Initiation Dose 30 μg/kg/h (N=5)
Severe intradialytic hypertension (Cardiac disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No